CLINICAL TRIAL: NCT06752707
Title: MiGo Tracker: Seamless Remote Therapeutic Monitoring of Exercise Adherence After Stroke
Brief Title: MiGo Tracker Remote Monitoring of Home Exercise After Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flint Rehabilitation Devices, LLC (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Rancho Research Institute, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R44AG090216-01 (NIH); R44AG090216-01 (NIH)
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Subacute Stroke
Keywords: Remote Therapeutic Monitoring; Stroke; Home Exercise Therapy; MiGo Tracker
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MiGo Tracker enabled RTM Program (Experimental): Participants will be provided a MiGo Tracker device which will log all home exercise sessions and uploaded to the MiGo-RTM dashboard. The supervising study therapist will conduct weekly phone calls with each participant where they review exercise metrics and assist with any barriers or issues.
  Interventions: Device: MiGo Tracker
- Conventional Standard of Care (Active Comparator): Participants will be assigned a home exercise regimen designed by a study therapist based on the individual participant's specific goals and abilities.
  Interventions: Other: Conventional home exercise program

INTERVENTIONS:
Device: MiGo Tracker — Perform home exercise sessions while wearing MiGo Tracker device that logs exercise data.
  Arms: MiGo Tracker enabled RTM Program
Other: Conventional home exercise program — Exercise following printed sheets or booklet
  Arms: Conventional Standard of Care

SUMMARY:
This project will determine the safety and effectiveness of a MiGo Tracker RTM program in a randomized controlled trial with individuals with subacute stroke (N=50). Participants will be randomly assigned to either the MiGo Tracker RTM program (intervention group) or prescription of home exercises with no monitoring (usual care/control group). All participants will still receive usual post-stroke care, including outpatient rehabilitation. The main question this study aims to answer is: Does a MiGo Tracker RTM program lead to significantly greater motor recovery at three-months post stroke than the usual care group. If successful, MiGo Tracker will lead to increased home exercise adherence and improved health outcomes for thousands of individuals following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Experienced one or more strokes less than one month (30 days) prior
* Upper Extremity Fugl-Meyer Score > 5 and <= 55 out of 66
* Absence of moderate to severe pain (<= 4 on the 10 point visual-analog pain scale)

Exclusion Criteria:

* age <18 years old
* Unable to follow 2-step commands
* Other neurological diagnosis (e.g. Parkinson's Disease)
* Other severe concurrent medical conditions that may prevent the participants from completing the 3-month study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Upper Extremity Fugl-Meyer from Baseline | Baseline and 3 months post stroke
  The Fugl-Meyer Assessment - Upper Extremity (FMA-UE) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, sensation, balance, joint range of motion and joint pain in patients with post-stroke hemiplegia. A standardized assessment of arm impairment based on scores of 0-2 on 33 different tasks. Minimum value = 0, maximum value = 66, higher scores = better outcome

SECONDARY OUTCOMES:
Change in Action Research Arm Test from Baseline | Baseline and 3 months post stroke
  The Action Research Arm Test (ARAT) is a 19-item measure aimed at assessing functional performance of the upper extremity through observational means. The ARAT is a 19 item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). Performance on each item is rated on a 4-point ordinal scale ranging from:
  (3) Performs test normally (2) Completes test, but takes abnormally long or has great difficulty
  (1) Performs test partially (0) Can perform no part of test
Change in Box and Blocks from Baseline | Baseline and 3 months post stroke
  The Box and Block Test assesses unilateral gross manual dexterity. The test is scored by counting the number of blocks carried over the partition from one compartment to the other during the one-minute trial period.
Change in Motor Activity Log from Baseline | Baseline and 3 months post stroke
  The MAL is a semi-structured interview to assess arm function. Individuals are asked to rate Quality of Movement (QOM) and Amount of Movement (AOM) during 30 daily functional tasks. Items scored on a 6-point ordinal scale.
  Scoring on Amount of Use Scale: 0) The weaker arm was not sued at all for that activity (never) 1) very rarely 2) rarely 3) half pre-stroke 4)3/4 pre-stroke 5) normal. Quality of Movement Scale: 0) The weaker arm was not used at all for that activity (never) 1) very poor 2) poor 3) fair 4) almost normal 5) normal
Change in Modified Ashworth Spasticity Scale from Baseline | Baseline and 3 months post stroke
  MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0-4 ordinal scale. The grade is assigned by moving a joint/muscle through a high velocity quick stretch. A score of 1 indicates no resistance, and 5 indicates rigidity.
Change in Visual Analog Pain Scale from Baseline | Baseline and 3 months post stroke
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10cm line that represents a continuum between "no pain" and "worst pain".

CONTACTS AND LOCATIONS:
Locations (1):
- Rancho Research Institute, Inc, Downey, California, United States

IPD SHARING:
Plan to Share IPD: Undecided